CLINICAL TRIAL: NCT07016971
Title: A Pilot Study to Evaluate the Feasibility, Safety, and Efficacy of Cannabigerol/Cannabidiol Oil for Chemotherapy-Induced Peripheral Neuropathy
Brief Title: CBG/CBD Oil for Chemotherapy-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Wesley Raup-Konsavage, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSCI-24-119
Record Dates: First submitted 2025-05-30; First posted 2025-06-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBG/CBD Oil Treatment Arm (Experimental): This is a single-arm, open-label study in which all participants will receive the intervention of CBG/CBD oil treatment. Participants will be administered sublingual CBG/CBD oil for 12 weeks. The initial dose will be 0.5 mL (17 mg of cannabinoids) twice daily for the first week, followed by 1 mL (33 mg of cannabinoids) twice daily for the remaining 11 weeks. The treatment period is divided into three 4-week cycles. Weekly remote safety phone calls will be conducted, and follow-up phone calls will take place one month after the last dose to monitor safety. The primary goals are to evaluate the safety, tolerability, and feasibility of the CBG/CBD oil, while secondary goals include assessing changes in CIPN symptoms, physical function, mental health, pharmacological tolerance, and adherence to the treatment.
  Interventions: Drug: CBG/CBD Oil

INTERVENTIONS:
Drug: CBG/CBD Oil — Participants will receive a commercially available high CBG/CBD hemp extract oil that also contains small amounts of cannabichromene (CBC). The product is formulated as a sublingual oil and administered twice daily. Participants will take 0.5 mL of the oil sublingually twice daily during the first week, followed by 1 mL sublingually twice daily for the remaining 11 weeks. The oil has a defined and independently verified cannabinoid and terpene profile and is marketed as a dietary supplement.

SUMMARY:
The goal of this clinical trial is to learn if a commercially available cannabigerol (CBG)/cannabidiol (CBD) oil is safe, feasible to use, and can help reduce symptoms of chemotherapy-induced peripheral neuropathy (CIPN) in adults who have completed platinum-based chemotherapy for gastrointestinal cancers. The main questions it aims to answer are:

Is CBG/CBD oil safe and well-tolerated over a 12-week treatment period?

Can participants with CIPN use CBG/CBD oil consistently as part of their care?

Does CBG/CBD oil help reduce pain, numbness, or other symptoms of CIPN?

Participants will:

Take CBG/CBD oil under the tongue (sublingually) twice daily for 12 weeks

Complete regular symptom assessments and functional tests during study visits

Provide blood samples for cannabinoid and metabolite level testing

DETAILED DESCRIPTION:
This pilot clinical trial is designed to evaluate the safety, feasibility, and preliminary efficacy of a commercially available cannabigerol (CBG)/cannabidiol (CBD) oil in treating chemotherapy-induced peripheral neuropathy (CIPN) in adult patients who have completed platinum-based chemotherapy for gastrointestinal malignancies. The study is based on preclinical findings from Dr. Wesley Raup-Konsavage's laboratory, which showed that CBG and CBD reduced neuropathic pain in animal models of CIPN. This clinical trial seeks to translate these findings into a patient population with persistent CIPN symptoms.

The study intervention uses a high-CBG/CBD hemp oil extract that is marketed as a dietary supplement and contains a verified profile of cannabinoids and terpenes. The formulation also includes small amounts of cannabichromene (CBC), which may contribute to analgesic effects via the "entourage effect." Subjects will administer 0.5 mL sublingually twice daily during the first week, followed by 1 mL sublingually twice daily for the remaining 11 weeks of the 12-week treatment period.

The treatment period is divided into three 4-week cycles to structure visit scheduling and assessments. The study will collect data on symptom changes, physical function, mental health, tolerability, and cannabinoid levels over time.

Primary objectives include evaluating the safety and tolerability of CBG/CBD oil and the feasibility of its use in this patient population. Secondary objectives include measuring changes in CIPN symptoms, physical and mental function, adherence, pharmacological tolerance, and circulating cannabinoid/metabolite levels.

The study addresses an urgent need for effective treatments for CIPN, as current therapies (e.g., duloxetine, gabapentin, NSAIDs) are often inadequate and poorly tolerated. By assessing a hemp extract rather than a purified compound, this study also explores the broader applicability and real-world relevance of cannabinoid-based supplements for supportive cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years or older.
* Patients with grade 1 or greater CIPN symptoms, such as neuropathic pain, paresthesia, or muscle weakness, persisting for more than 2 weeks as defined by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 5.
* Patients who have completed platinum-based chemotherapy for colorectal carcinoma, biliary tract carcinoma, pancreatic carcinoma, esophageal carcinoma, gastric carcinoma, or small intestinal carcinoma within the past 2 years.
* Patients currently taking any treatment for CIPN must discontinue such treatments at least 2 weeks prior to enrollment.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (To be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 1 months after the last dose of protocol therapy. Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).
* Patients from Penn State Health.

Exclusion Criteria:

* Patients under the age of 21 years.
* Patients with a history of preexisting neuropathy prior to chemotherapy.
* Pregnant and nursing women.
* Patients with hypertension that, in the investigator's judgement, is uncontrolled despite the use of anti-hypertensives, or with hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <60 mmHg).
* History of or active arterial thromboembolic event (e.g. stroke, myocardial infarction).
* Patients who have used an investigational drug within 30 days prior to the screening visit or are currently participating in another interventional investigational study.
* Patients who have liver function tests AST/ALT > 3 times above the upper limits of normal (ULN) in the past year.
* Patients who have suicidal ideation or uncontrolled depression within the past year.
* Patients with known sensitivity to any components of CBG/CBD hemp extract.
* Patients with known sensitivity to coconut oil.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of CBG/CBD Oil | Through study completion (12 weeks)
  Evaluated by the incidence and severity of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. The NCI CTCAE v5.0 grades adverse events on a scale from 1 to 5, where:
  Grade 1: Mild; asymptomatic or mild symptoms. Grade 2: Moderate; minimal, local, or noninvasive intervention indicated. Grade 3: Severe or medically significant but not immediately life-threatening. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to adverse event. Minimum value: Grade 1 (mild). Maximum value: Grade 5 (death). Interpretation: Higher grades indicate worse outcomes (more severe adverse events).
  Focus will be on toxicities of grade 2 or higher throughout the 12-week treatment period (Cycles 1-3).
Feasibility of Treatment with CBG/CBD Oil | Week 4 (End of Cycle 1)
  Defined as the percentage of participants who complete Cycle 1 (Weeks 1-4) of study participation, including all required visits, assessments, and adherence to CBG/CBD oil dosing.

SECONDARY OUTCOMES:
Changes in CIPN Symptoms | At the end of Cycle 1 (Week 4), Cycle 2 (Week 8), and Cycle 3 (Week 12); each cycle is 28 days.
  The PNQ grades the severity of chemotherapy-induced peripheral neuropathy (CIPN) symptoms on a scale from 0 to 4, where:
  0: No neuropathy.
  1. Mild neuropathy; does not interfere with daily activities.
  2. Moderate neuropathy; some interference with daily activities.
  3. Severe neuropathy; significant interference with daily activities.
  4. Disabling neuropathy; prevents daily activities. Minimum value: 0 (no neuropathy). Maximum value: 4 (disabling neuropathy). Interpretation: Higher scores indicate worse outcomes (more severe neuropathy symptoms).
  Symptoms will be assessed for changes in sensory and motor disturbances and their impact on daily activities.
Changes in Physical Function | At the end of Cycle 1 (Week 4), Cycle 2 (Week 8), and Cycle 3 (Week 12); each cycle is 28 days.
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 20a. This scale assesses the impact of muscle weakness associated with chemotherapy-induced peripheral neuropathy (CIPN) on daily activities. The PROMIS Physical Function Short Form 20a consists of 20 items, with responses scored from 1 to 5:
  1: Unable to do or severe limitation. 5: No difficulty or limitation. Minimum value: 20 (indicating severe limitation across all items). Maximum value: 100 (indicating no limitation across all items). Interpretation: Higher scores indicate better outcomes (better physical function).
  Physical function will be assessed by comparing baseline scores to those collected at the end of each cycle.
Changes in Mental Health Scores | At the end of Cycle 1 (Week 4), Cycle 2 (Week 8), and Cycle 3 (Week 12); each cycle is 28 days.
  Assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress - Anxiety Short Form 8a and PROMIS Cognitive Function - Short Form 8a.
  Anxiety Short Form 8a: 8 items, scored 1 (never) to 5 (always); T-scores range from ~37.1 (minimal anxiety) to ~83.1 (severe anxiety). Higher T-scores indicate worse outcomes.
  Cognitive Function Short Form 8a: 8 items, scored 1 (poor function) to 5 (good function); T-scores range from ~25.0 (poor) to ~75.0 (excellent). Higher T-scores indicate better outcomes.
  Changes in T-scores from baseline to end of each cycle.
Pharmacological Tolerance to CBG/CBD Oil | At the end of Cycle 1 (Week 4), Cycle 2 (Week 8), and Cycle 3 (Week 12); each cycle is 28 days.
  Measured by changes in Patient Neurotoxicity Questionnaire (PNQ) scores, assessing the decrease in the effectiveness of CBG/CBD oil treatment for chemotherapy-induced peripheral neuropathy (CIPN) symptoms. The PNQ grades the severity of sensory and motor disturbances on a scale from 0 to 4, where:
  0: No neuropathy.
  1. Mild neuropathy; does not interfere with daily activities.
  2. Moderate neuropathy; some interference with daily activities.
  3. Severe neuropathy; significant interference with daily activities.
  4. Disabling neuropathy; prevents daily activities. Minimum value: 0 (no neuropathy). Maximum value: 4 (disabling neuropathy). Interpretation: Higher scores indicate worse outcomes (more severe neuropathy symptoms, suggesting decreased treatment effectiveness).
  Changes in PNQ scores will be evaluated by comparing baseline scores to those collected at the end of each cycle to assess potential pharmacological tolerance.
Changes in Circulating Cannabinoids and CBD Metabolites | At the end of Cycle 2 (Week 8); each cycle is 28 days.
  Measured as the difference in plasma concentrations of cannabinoids and CBD metabolites (e.g., CBG, CBD, and their metabolites) from baseline to the end of Cycle 2. Plasma levels will be quantified using validated analytical methods (liquid chromatography-mass spectrometry).
Adherence to CBG/CBD Oil Treatment | During Cycle 1 (Weeks 1-4), Cycle 2 (Weeks 5-8), and Cycle 3 (Weeks 9-12); each cycle is 28 days.
  Defined as the proportion of prescribed CBG/CBD oil doses taken per cycle. Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Medication Adherence Scale and patient drug diaries.
  PROMIS Medication Adherence Scale: Items scored 1 (never) to 5 (always); T-scores range from ~30.0 (poor adherence) to ~70.0 (excellent adherence). Higher T-scores indicate better outcomes.
  Drug Diaries: Record daily doses to calculate proportion taken. Adherence assessed by combining T-scores and diary data per cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Yee, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States